CLINICAL TRIAL: NCT00140296
Title: Using the Healthcare Visit to Improve Contraceptive Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCCDPHP-TS-0768
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Pregnancy; Chlamydia
MeSH Terms: conditions — Chlamydia Infections

INTERVENTIONS:
Behavioral: Contraceptive counseling

SUMMARY:
Consistent and correct use of an effective contraceptive method is a primary determinant in preventing pregnancy. Unfortunately, only a minority of healthcare providers adequately address women's contraceptive needs. We have developed a standardized behavioral-based contraceptive counseling model that can be used by providers and other clinic staff to address this limitation. The model, ESP, is an adaptation of motivational interviewing and involves: Exploring discrepancies between pregnancy intention and contraceptive use and between risk of STDs and condom use; Sharing information; and Promoting behaviors to reduce risk.

Study question: Does ESP counseling lead to an increase in consistency and effectiveness of contraceptive use among women at risk of unintended pregnancy?

Methods: Randomized controlled trial of 747 women, ages 16-44, at self-identified risk of unintended pregnancy enrolled from March 2003 to September 2004 at healthcare settings in North Carolina. Intervention participants received individualized ESP counseling from a health educator to address barriers to effective and consistent contraceptive use. Risk reduction steps were negotiated. Pregnancy, Chlamydia infection and contraceptive use were assessed at baseline and follow-up. "Highly effective" contraceptive use was defined as a combination of effectiveness and consistency. Women in the control arm received general preventive health counseling (e.g., smoking and exercise). Differences between the study arms at 12-months may illustrate the longer term influence of the intervention.

DETAILED DESCRIPTION:
Consistent and correct use of an effective contraceptive method is a primary determinant in preventing pregnancy. Unfortunately, only a minority of healthcare providers adequately address women's contraceptive needs. We have developed a standardized behavioral-based contraceptive counseling model that can be used by providers and other clinic staff to address this limitation. The model, ESP, is an adaptation of motivational interviewing and involves: Exploring discrepancies between pregnancy intention and contraceptive use and between risk of STDs and condom use; Sharing information; and Promoting behaviors to reduce risk.

Study question: Does ESP counseling lead to an increase in consistency and effectiveness of contraceptive use among women at risk of unintended pregnancy?

Methods: Randomized controlled trial of 747 women, ages 16-44, at self-identified risk of unintended pregnancy enrolled from March 2003 to September 2004 at healthcare settings in North Carolina. Intervention participants received individualized ESP counseling from a health educator to address barriers to effective and consistent contraceptive use. Risk reduction steps were negotiated. Pregnancy, Chlamydia infection and contraceptive use were assessed at baseline and follow-up. "Highly effective" contraceptive use was defined as a combination of effectiveness and consistency. Women in the control arm received general preventive health counseling (e.g., smoking and exercise). Differences between the study arms at 12-months may illustrate the longer term influence of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16-44
* English-speaking
* Do not wish to be pregnant or unsure of pregnancy intention
* Have an appointment for non-acute care
* Currently using no method of contraception, inconsistent use of methods, pills, condoms, diaphragms, periodic abstinence, or methods associated with higher pregnancy rates
* Ability to read at least at 8th grade level
* Willing to participate in follow-up visits at 2, 8, and 12 months
* Able to be contacted by telephone

Exclusion Criteria:

* Women less than 16 or greater than 44 years
* Women who are sterilized, or whose partners are sterilized or who use the IUD for contraception
* Appointments for acute care
* Non-English speaking
* Inability to read at or above 8th grade level
* Pregnant at time of enrollment
* Lack of ability for telephone contact

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 747
Dates: Start 2003-03; Study Completion 2005-09

PRIMARY OUTCOMES:
Contraceptive use
Chlamydia infection
Pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Petersen, MD, MPH, Principal Investigator — University of North Carolina
Locations (1):
- Center for Women's Health Research, Universoty of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Petersen R, Payne P, Albright J, Holland H, Cabral R, Curtis KM. Applying motivational interviewing to contraceptive counseling: ESP for clinicians. Contraception. 2004 Mar;69(3):213-7. doi: 10.1016/j.contraception.2003.10.007. PMID 14969669